CLINICAL TRIAL: NCT06491121
Title: Technology Supported High Intensity Training in Chronic Low Back Pain: the Techno-HIT Trial
Acronym: TECHNO-HIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Annick Timmermans, Professor Doctor, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: T000822N
Record Dates: First submitted 2024-05-29; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Chronic Low-back Pain; Exercise Therapy; Telerehabilitation
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: A double blind (outcome assessor & statistical analysis) three-armed multicentre RCT will be conducted. This RCT will adhere to Good Clinical Practice (GCP) regulations.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TECHNO-HIT group (Experimental): Technology supported High Intensity Training
  Interventions: Other: Technology supported High Intensity Training
- HIT group (Experimental): High Intensity Training
  Interventions: Other: High Intensity Training
- MIT group (Active Comparator): Moderate Intensity Training
  Interventions: Other: Moderate Intensity Training

INTERVENTIONS:
Other: Technology supported High Intensity Training — patients will perform a 12-week HIT program comprising of 1,5h exercise therapy sessions twice a week. The program is a combination of cardiorespiratory interval, general resistance, and core muscle strength training, all at high intensity. phase 2 is a similar 12-week HIT program at home, supported by a smartphone application
  Arms: TECHNO-HIT group
Other: Moderate Intensity Training — patients will perform a 12-week MIT program comprising of 1,5h exercise therapy sessions twice a week. The program is a combination of cardiorespiratory continuous load, general resistance and core muscle training, all at moderate intensity. Phase 2 is a similar 12-week MIT program at home with an exercise program on paper.
  Arms: MIT group
Other: High Intensity Training — patients will perform a 12-week HIT program comprising of 1,5h exercise therapy sessions twice a week. The program is a combination of cardiorespiratory interval, general resistance, and core muscle strength training, all at high intensity. phase 2 is a similar 12-week HIT program at home with an exercise program on paper.
  Arms: HIT group

SUMMARY:
Chronic low back pain (CLBP) is one of the most common chronic musculoskeletal disorder worldwide and is responsible for the highest levels of disability of all diseases. All state-of-the-art guidelines recommend implementing exercise therapy (ET) in CLBP management. Researchers have shown that a novel ET modality, namely high intensity training (HIT), can be valuable. A clinical evaluation study in a larger spectrum of persons with CLBP in a rehabilitation centre setting is essential. Thereby, technology might support HIT.

The primary goal of this clinical trial is to evaluate the short- and long-term effectiveness of a time contingent individualized High intensity training (HIT) protocol on disability compared to moderate intensity training (MIT) in persons with severely disabling chronic low back pain (CLBP). Secondary goals entail 1) evaluating short- and long-term effectiveness of HIT on psychosocial correlates, central pain processing, and broad physical fitness, 2) investigating additional effects of (prolonged) HIT at home, 3) investigating added value of technology through a mobile (smartphone) and dashboard (computer) application that offers support during home training, 4) evaluating cost-effectiveness of (technology supported) HIT compared to MIT. The main research question[s] (RQ) it aims to answer are:

* RQ1: To what extent is HIT effective on the short- and long term to improve disability in persons with severely disabling CLBP compared to MIT as used in usual care?
* RQ2a: To what extent does HIT have a short- and/or long-term effect on central pain processing and psychosocial correlates in persons with severely disabling CLBP?
* RQ2b:To what extent does HIT have a short- and/or long-term effect on outcomes related to broad physical fitness in persons with severely disabling CLBP?
* RQ3a: To what extent does prolonged (technology-supported) HIT at home provide additional training effects in persons with severely disabling CLBP?
* RQ3b:To what extent does a mobile application that offers support for HIT at home provide added value for treatment outcomes of persons with severely disabling CLBP?
* RQ3c:To what extent is the techno-HIT application usable and qualitative (assessed by SUS and uMARS) as a therapeutic support mechanism, as evaluated by persons with severely disabling CLBP?
* RQ4: To what extent is HIT or HIT supported by a mobile application cost effective compared to MIT for patients with severely disabling CLBP?

DETAILED DESCRIPTION:
This RCT includes a total sample size of n=168 persons with chronic low back pain (CLBP) randomly divided into three groups of each 56 participants (Group 1: 'TechnoHIT'; Group 2: 'HIT'; Group 3: 'MIT'). For each group, the trial involves a 24-week exercise intervention with a total of 52 rehabilitation sessions (4 educational sessions in the biopsychosocial program in the first two weeks and two physical therapy sessions each week (n=48 in total)) in three phases (2 therapy phases and 1 follow- up phase). The first therapy phase consists of 12 weeks and is performed in the hospitals (Jessa and UZA) under supervision of PhD-students (with a physiotherapy background) that are members of the FWO TECHNOHIT consortium and clinical study assistants (with a physiotherapy background). The second therapy phase consists of 12 weeks and is performed in the home setting of the participant. The follow-up phase only consists of advice towards continuation of physical activity and app logging or no contact based on group randomization. The first follow-up visit is planned directly after the last treatment session in the hospital. The second follow-up visit will take place 3 months after the last treatment session, shortly after the last at-home session. The last two follow-up visits will take place 6 and 18 months after the last at-home session.

Patients with CLBP who present themselves at UZA/Jessa for consultation and start-up of a rehabilitation program (i.e. within the Belgian reimbursement system for medical treatments defined as a 'K60 programma: Ambulante multidisciplinaire revalidatiezitting met een minimumduur van 120 minuten voor een wervelzuilaandoening') who ought to be eligible for the study by the physician (=who meet the inclusion criteria), will be informed about this study by the physician. If they are interested, a study flyer and an approval form for further contact will be issued by the physician. The form is signed by the patient and returned. The researchers will contact the potential participant within a period of two to seven days, answer initial questions, review the inclusion criteria, and provide the informed consent (online/hard copy according to the preference of the potential participant). Patients who sign and return the informed consent within two weeks will be contacted for possible enrolment.

This study will start recruitment in January 2024 and have an active intervention phase of three years. The end of the recruitment phase is therefore planned around January 2027. After the recruitment phase, a period of six months is reserved for final data analysis and scientific publication writing. The total duration of this study is therefore 3.5 years (the end of the study is expected around August 2027).

Pre-phase: biopsychosocial education program (4 sessions, T-1-T0):

Four sessions with educational content (60 min./session, 2x/week) will be organized at the hospitals at the start of the intervention for all groups. This educational content relates to a) pain education/dealing with pain, b) ergonomics, c) activity management and optimizing the working and social environment, and d) neurophysiology of pain. These sessions will be provided by the PhD students. The content of this education program is based on scientific research and publications on patient education from renowned organizations such as retrainpain.org and pain in motion and on extensive work previously done by members of the consortium. The content will be standardized between the test centers UZA and Jessa.

Phase 1: intervention at the hospital facility (24 sessions, week 1-12, T0-T1) The three groups will follow a 12-week training program in which a time contingent approach is used as proposed by recent clinical practice guidelines. To limit performance bias, each group will train separately and will not be able to evaluate differences between the therapies.

Group 1 ('TechnoHIT') and group 2 ('HIT') - These groups will perform 1,5h exercise therapy sessions twice a week comprising of a combination of cardiorespiratory interval, general resistance, and core muscle strength training, all at high intensity, according to a previously published protocol by our research group. Briefly, cardiorespiratory training consists of an interval protocol on a cycle ergo-meter consisting of five one-minute 100% VO2max workload bouts, separated by one minute of active rest at 50% VO2max workload. 100% VO2max bouts increase every two sessions by 10''. Active rest remains stable. This protocol is repeated from session 13 to 24 with an updated workload (+5% WMax). General resistance training consists of three upper body and three lower body exercises executed on fitness equipment performed at 80% of the one repetition maximum. Core muscle strength training consists of six static core exercises and related progressions. Exercises were chosen in function of their ability to load the core muscles at an intensity of >60% of the maximum voluntary contraction.

Group 3 ('MIT', control group) - This group will perform 1,5h exercise therapy sessions twice a week of cardiorespiratory continuous load, general resistance and core muscle training, all at moderate intensity, according to a previously published protocol by our research team. Briefly, cardiorespiratory training consists of a continuous training protocol on a cycle ergometer. Participants start with 14 minutes of cycling (90 repetitions per minute at 60%VO2max workload). Duration will be increased every two sessions with 1'40'' up to 22'40''. This protocol is repeated from session 13 to 24 with an updated workload (+5% WMax). General resistance training is identical to the protocol described in 'HIT' with the exception of the exercise intensity (exercises are performed here at 60% of 1RM). Core muscle strength training is identical to the protocol described in 'HIT' with the exception of the exercise intensity. Participants perform one set of ten repetitions of a ten second static hold. Exercises are made more difficult when they were executed with a stable core posture for the indicated time by increasing the time of the static hold each six sessions.

Phase 2: intervention at home (24 sessions, week 13-24, T1-T2) The three groups will follow a comparable 12-week training program as phase 1 but in their home setting. The participants of group 1 will be supported by a mobile application on their phone. The participants of group 1 & 2 will be provided with a fitness bike, a smartwatch (Polar M200), and training mat during the execution of this phase. Sessions missed by the participants because of adverse events (e.g., acute increase of low back pain, acute musculoskeletal issues due to exercises) will be registered.

Group 1 ('TECHNO-HIT') - Participants in this group receive an exercise schedule via the TechnoHIT mobile application, a home trainer (E50, Tunturi Fitness), a heartrate sensor (H10, Polara) and smartwatch (Ignite, Polar), and a training mat for the duration of this phase. They are asked to perform a 60 min. home program twice a week containing cardiorespiratory and core muscle strength training, both at high intensity (HIT protocol methods are equal to those in Phase 1). The training sessions of these patients are guided by the mobile application. The user reports performes exercises in the mobile application, that keeps track of their progress, calculates compliance with the program and gives motivational feedback based on the patient's performance and adherence.

Group 2 ('HIT') - Participants in this group receive an exercise schedule on paper, a home trainer (i.e. fitness bike) and a training mat for the duration of this phase. They are asked to perform a one-hour home program twice a week containing cardiorespiratory and core muscle strength training, both at high intensity. They also receive a diary to log their training sessions.

Group 3 ('MIT', control group) - Participants in this group receive an exercise schedule on paper. They are asked to perform a one-hour home program twice a week containing cardiorespiratory and core muscle training, both at moderate intensity. They also receive a diary to log their training sessions. As we decided not to provide a bicycle and exercise mat in order to match the "therapy as usual" setting, cardiorespiratory training in this phase will be based on a brisk walking modality performed at the same moderate exercise intensity and matched for training volume.

The Techno-HIT home-training system consists of the following components and main functionalities:

* a mobile application for the patients at home (to receive the HIT training program, to schedule the training in sessions over the week, to receive reminders and notifications, to see the overall HIT training program or get more details on exercises and performed sessions, to have access to exercise instructions, to get guidance by the app while performing the exercises, to get motivational feedback after performing the exercise and reporting the status, to get feedback about progress and adherence, to select a strategy to improve the adherence, to report a variety of activities beyond the HIT program, etc.);
* a dashboard application for the physiotherapists / researchers (to see an overview of notifications about the patient's training status, to search through patient files and notifications, to manage patient groups, to provide the info on the HIT training, to update exercise parameters, to follow-up on the patients' progress and view aggregated visual representations of progress, to send hints to the patients, to follow system suggestions for a progression or regression, to give feedback to patients). Some functionalities are "admin" functionalities and require an authorized account (e.g. to create new patient files, to manage caregiver accounts, etc.).

Participants perform two assessments at baseline (T-1: PRE before psychosocial education & T0: PRE after psychosocial education), and 4 longitudinal assessment (T1: MID after a 12-week program in-hospital, T2: POST after a 12-week program at home, T3: POST 6 month follow-up, T4: POST 18 month follow-up) consisting of both physical testings and filling in health and disease related questionnaires. At T-1, the assessments have a duration of approximately 2 hours (90min questionnaires + 30min QST measurements). During this assessment, sociodemographic data of the participant will also be collected. At T0, physical assessments will be added, aswell as additional questionnaires. T0 will have a duration of approximately 3 hours. At T1, T2, T3 and T4, additional questionnaires will be added, increasing the duration to 3 hours and 40 minutes.

A rater cross-over assessment protocol will be used to ensure blinding of assessors. All assessments are carried out by trained PhD-students and postdoctoral researchers that are part of the FWO Techno-HIT Trial project in the specialized movement and pain assessment labs of REVAL, UHasselt and MOVANT, UAntwerpen. (see section outcomes for detailed information on the depicted outcome measures)

All data is treated confidentially and encrypted during the execution of the tests ('HIT-TECH', followed by a timing letter/number (T-1 =A, T0=0, T1=1, T2=2, T3=3, T4=4) and a sequence number (01 to 15)). To associate the data with the subjects during data analysis, a subject identification list (0-15, randomized) is used. The identification and key of the code is monitored by an independent researcher who is not involved in the research. All data collected is stored in the Google Drive (UHasselt)/Microsoft Teams (UAntwerp) file stream and only members of the research team with a university account and password can access the source data. Source data is kept for 25 years in accordance with GCP standards for reuse or for results validation.

ELIGIBILITY:
Inclusion Criteria:

* speak Dutch
* be 18 to 65 years old
* have nonspecific CLBP defined as chronic primary musculoskeletal pain (ICD-11: MG30.011) in the low back persisting for at least 12 weeks12, whereby fluctuations in pain can be present and pain can be alternated by remission phases. Furthermore, regarding the specification of 'severity', only participants with a profile consisting of a score of >20% on the Modified Oswestry disability Index (i.e. 'moderate disability') will be included.
* have and make use of a working iOS/Android smartphone

Exclusion Criteria:

* when they have had spinal fusion surgery
* when they have a musculoskeletal and/or chronic disorder aside from CLBP that could affect the correct execution of the therapy program or evaluation of the outcomes
* when they have severe comorbidities (e.g., paresis or sensory disturbances by neurological causes, diabetes mellitus, rheumatoid arthritis)
* when they are pregnant
* when they have ongoing compensation claims
* when they are not able to attend regular therapy appointments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Modified Oswestry Disability Index (MODI) questionnaire - Time necessary for completion: 5 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  This questionnaire is used to evaluate disability and consists of ten items scored on a five-point scale (0-5) whereby zero means minimal disability and five means very severe disability. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Modified Oswestry Disability Index (MODI) questionnaire - Time necessary for completion: 5 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire is used to evaluate disability and consists of ten items scored on a five-point scale (0-5) whereby zero means minimal disability and five means very severe disability. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Modified Oswestry Disability Index (MODI) questionnaire - Time necessary for completion: 5 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire is used to evaluate disability and consists of ten items scored on a five-point scale (0-5) whereby zero means minimal disability and five means very severe disability. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Modified Oswestry Disability Index (MODI) questionnaire - Time necessary for completion: 5 min | T2: POST (After completing the 12-week protocol at home)
  This questionnaire is used to evaluate disability and consists of ten items scored on a five-point scale (0-5) whereby zero means minimal disability and five means very severe disability. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Modified Oswestry Disability Index (MODI) questionnaire - Time necessary for completion: 5 min | T3: POST (6 months follow-up)
  This questionnaire is used to evaluate disability and consists of ten items scored on a five-point scale (0-5) whereby zero means minimal disability and five means very severe disability. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Modified Oswestry Disability Index (MODI) questionnaire - Time necessary for completion: 5 min | T4: POST (18 months follow-up)
  This questionnaire is used to evaluate disability and consists of ten items scored on a five-point scale (0-5) whereby zero means minimal disability and five means very severe disability. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) - Time necessary for completion: 5 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  This questionnaire is used to evaluate (widespread) pain and consists of 9-items including a body chart to draw the pain region. A high score corresponds to more pain.
Brief Pain Inventory (BPI) - Time necessary for completion: 5 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire is used to evaluate (widespread) pain and consists of 9-items including a body chart to draw the pain region. A high score corresponds to more pain.
Brief Pain Inventory (BPI) - Time necessary for completion: 5 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire is used to evaluate (widespread) pain and consists of 9-items including a body chart to draw the pain region. A high score corresponds to more pain.
Brief Pain Inventory (BPI) - Time necessary for completion: 5 min | T2: POST (After completing the 12-week protocol at home)
  This questionnaire is used to evaluate (widespread) pain and consists of 9-items including a body chart to draw the pain region. A high score corresponds to more pain.
Brief Pain Inventory (BPI) - Time necessary for completion: 5 min | T3: POST (6 months follow-up)
  This questionnaire is used to evaluate (widespread) pain and consists of 9-items including a body chart to draw the pain region. A high score corresponds to more pain.
Brief Pain Inventory (BPI) - Time necessary for completion: 5 min | T4: POST (18 months follow-up)
  This questionnaire is used to evaluate (widespread) pain and consists of 9-items including a body chart to draw the pain region. A high score corresponds to more pain.
Quantitative sensory testing (QST) thermal stimuli - Time necessary for completion: 30 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  QST will be used to examine nociceptive processing of pain by applying various thermal stimuli at affected and remote sites. Advanced thermal stimulation will be assessed with the TSA II (Medoc), including thermal pain thresholds, temporal summation, and conditioned pain modulation (CPM). CPM will be examined to evaluate the endogenous analgesic system, by examining the change in pain perceived in one body region (test stimulation) as a result of pain induced in another body region (conditioned stimulation).
Quantitative sensory testing (QST) thermal stimuli - Time necessary for completion: 30 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  QST will be used to examine nociceptive processing of pain by applying various thermal stimuli at affected and remote sites. Advanced thermal stimulation will be assessed with the TSA II (Medoc), including thermal pain thresholds, temporal summation, and conditioned pain modulation (CPM). CPM will be examined to evaluate the endogenous analgesic system, by examining the change in pain perceived in one body region (test stimulation) as a result of pain induced in another body region (conditioned stimulation).
Quantitative sensory testing (QST) thermal stimuli - Time necessary for completion: 30 min | T1: MID (After completing the 12-week protocol in hospital)
  QST will be used to examine nociceptive processing of pain by applying various thermal stimuli at affected and remote sites. Advanced thermal stimulation will be assessed with the TSA II (Medoc), including thermal pain thresholds, temporal summation, and conditioned pain modulation (CPM). CPM will be examined to evaluate the endogenous analgesic system, by examining the change in pain perceived in one body region (test stimulation) as a result of pain induced in another body region (conditioned stimulation).
Quantitative sensory testing (QST) thermal stimuli - Time necessary for completion: 30 min | T2: POST (After completing the 12-week protocol at home)
  QST will be used to examine nociceptive processing of pain by applying various thermal stimuli at affected and remote sites. Advanced thermal stimulation will be assessed with the TSA II (Medoc), including thermal pain thresholds, temporal summation, and conditioned pain modulation (CPM). CPM will be examined to evaluate the endogenous analgesic system, by examining the change in pain perceived in one body region (test stimulation) as a result of pain induced in another body region (conditioned stimulation).
Quantitative sensory testing (QST) thermal stimuli - Time necessary for completion: 30 min | T3: POST (6 months follow-up)
  QST will be used to examine nociceptive processing of pain by applying various thermal stimuli at affected and remote sites. Advanced thermal stimulation will be assessed with the TSA II (Medoc), including thermal pain thresholds, temporal summation, and conditioned pain modulation (CPM). CPM will be examined to evaluate the endogenous analgesic system, by examining the change in pain perceived in one body region (test stimulation) as a result of pain induced in another body region (conditioned stimulation).
Quantitative sensory testing (QST) thermal stimuli - Time necessary for completion: 30 min | T4: POST (18 months follow-up)
  QST will be used to examine nociceptive processing of pain by applying various thermal stimuli at affected and remote sites. Advanced thermal stimulation will be assessed with the TSA II (Medoc), including thermal pain thresholds, temporal summation, and conditioned pain modulation (CPM). CPM will be examined to evaluate the endogenous analgesic system, by examining the change in pain perceived in one body region (test stimulation) as a result of pain induced in another body region (conditioned stimulation).
Quantitative sensory testing (QST) Pinprick stimulator - Time necessary for completion: 5 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  Temporal summation will additionally be measured with the PinPrick-stimulator (MRC systems, 256mN) that will be repeatedly applied on the skin on the non-dominant forearm and the lower back, following a predefined standardized protocol. Wind-up ratio (WUR) is calculated comparing a single pinprick stimulus to trains of 10 pinprick stimuli. Stimuli are applied at a 1/s rate over a small area (1cm2) and the participant is asked to rate the pain on a scale of 0-100.
Quantitative sensory testing (QST) Pinprick stimulator - Time necessary for completion: 5 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  Temporal summation will additionally be measured with the PinPrick-stimulator (MRC systems, 256mN) that will be repeatedly applied on the skin on the non-dominant forearm and the lower back, following a predefined standardized protocol. Wind-up ratio (WUR) is calculated comparing a single pinprick stimulus to trains of 10 pinprick stimuli. Stimuli are applied at a 1/s rate over a small area (1cm2) and the participant is asked to rate the pain on a scale of 0-100.
Quantitative sensory testing (QST) Pinprick stimulator - Time necessary for completion: 5 min | T1: MID (After completing the 12-week protocol in hospital)
  Temporal summation will additionally be measured with the PinPrick-stimulator (MRC systems, 256mN) that will be repeatedly applied on the skin on the non-dominant forearm and the lower back, following a predefined standardized protocol. Wind-up ratio (WUR) is calculated comparing a single pinprick stimulus to trains of 10 pinprick stimuli. Stimuli are applied at a 1/s rate over a small area (1cm2) and the participant is asked to rate the pain on a scale of 0-100.
Quantitative sensory testing (QST) Pinprick stimulator - Time necessary for completion: 5 min | T2: POST (After completing the 12-week protocol at home)
  Temporal summation will additionally be measured with the PinPrick-stimulator (MRC systems, 256mN) that will be repeatedly applied on the skin on the non-dominant forearm and the lower back, following a predefined standardized protocol. Wind-up ratio (WUR) is calculated comparing a single pinprick stimulus to trains of 10 pinprick stimuli. Stimuli are applied at a 1/s rate over a small area (1cm2) and the participant is asked to rate the pain on a scale of 0-100.
Quantitative sensory testing (QST) Pinprick stimulator - Time necessary for completion: 5 min | T3: POST (6 months follow-up)
  Temporal summation will additionally be measured with the PinPrick-stimulator (MRC systems, 256mN) that will be repeatedly applied on the skin on the non-dominant forearm and the lower back, following a predefined standardized protocol. Wind-up ratio (WUR) is calculated comparing a single pinprick stimulus to trains of 10 pinprick stimuli. Stimuli are applied at a 1/s rate over a small area (1cm2) and the participant is asked to rate the pain on a scale of 0-100.
Quantitative sensory testing (QST) Pinprick stimulator - Time necessary for completion: 5 min | T4: POST (18 months follow-up)
  Temporal summation will additionally be measured with the PinPrick-stimulator (MRC systems, 256mN) that will be repeatedly applied on the skin on the non-dominant forearm and the lower back, following a predefined standardized protocol. Wind-up ratio (WUR) is calculated comparing a single pinprick stimulus to trains of 10 pinprick stimuli. Stimuli are applied at a 1/s rate over a small area (1cm2) and the participant is asked to rate the pain on a scale of 0-100.
Work Ability Index (WAI) - Time necessary for completion: 5 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  This questionnaire is used to evaluate self-perceived work ability in seven categories. The total score can range from 7 to 49 points with higher scores indicating better work ability
Work Ability Index (WAI) - Time necessary for completion: 5 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire is used to evaluate self-perceived work ability in seven categories. The total score can range from 7 to 49 points with higher scores indicating better work ability
Work Ability Index (WAI) - Time necessary for completion: 5 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire is used to evaluate self-perceived work ability in seven categories. The total score can range from 7 to 49 points with higher scores indicating better work ability
Work Ability Index (WAI) - Time necessary for completion: 5 min | T2: POST (After completing the 12-week protocol at home)
  This questionnaire is used to evaluate self-perceived work ability in seven categories. The total score can range from 7 to 49 points with higher scores indicating better work ability
Work Ability Index (WAI) - Time necessary for completion: 5 min | T3: POST (6 months follow-up)
  This questionnaire is used to evaluate self-perceived work ability in seven categories. The total score can range from 7 to 49 points with higher scores indicating better work ability
Work Ability Index (WAI) - Time necessary for completion: 5 min | T4: POST (18 months follow-up)
  This questionnaire is used to evaluate self-perceived work ability in seven categories. The total score can range from 7 to 49 points with higher scores indicating better work ability
Brief Resilience Scale (BRS-NL)- Time necessary for completion: 2 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  This questionnaire is used to evaluate the degree of individual resilience. The items of this self-report questionnaire are scored on a 5-point Likert scale. Possible scores are ranging from 1 to 5. A higher score corresponds to being more resilient than a lower score.
Brief Resilience Scale (BRS-NL)- Time necessary for completion: 2 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire is used to evaluate the degree of individual resilience. The items of this self-report questionnaire are scored on a 5-point Likert scale. Possible scores are ranging from 1 to 5. A higher score corresponds to being more resilient than a lower score.
Brief Resilience Scale (BRS-NL)- Time necessary for completion: 2 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire is used to evaluate the degree of individual resilience. The items of this self-report questionnaire are scored on a 5-point Likert scale. Possible scores are ranging from 1 to 5. A higher score corresponds to being more resilient than a lower score.
Brief Resilience Scale (BRS-NL)- Time necessary for completion: 2 min | T2: POST (After completing the 12-week protocol at home)
  This questionnaire is used to evaluate the degree of individual resilience. The items of this self-report questionnaire are scored on a 5-point Likert scale. Possible scores are ranging from 1 to 5. A higher score corresponds to being more resilient than a lower score.
Brief Resilience Scale (BRS-NL)- Time necessary for completion: 2 min | T3: POST (6 months follow-up)
  This questionnaire is used to evaluate the degree of individual resilience. The items of this self-report questionnaire are scored on a 5-point Likert scale. Possible scores are ranging from 1 to 5. A higher score corresponds to being more resilient than a lower score.
Brief Resilience Scale (BRS-NL) - Time necessary for completion: 2 min | T4: POST (18 months follow-up)
  This questionnaire is used to evaluate the degree of individual resilience. The items of this self-report questionnaire are scored on a 5-point Likert scale. Possible scores are ranging from 1 to 5. A higher score corresponds to being more resilient than a lower score.
Tampa Scale for Kinesiophobia (TSK) - Time necessary for completion: 10 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  This questionnaire is used to evaluate fear of movement and fear of (re)injury on a 4-point Likert scale ranging from "strongly disagree" to "strongly agree". Items 4, 8, 12 and 16 are inversely phrased. A higher score indicates higher levels of kinesiophobia.
Tampa Scale for Kinesiophobia (TSK) - Time necessary for completion: 10 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire is used to evaluate fear of movement and fear of (re)injury on a 4-point Likert scale ranging from "strongly disagree" to "strongly agree". Items 4, 8, 12 and 16 are inversely phrased. A higher score indicates higher levels of kinesiophobia.
Tampa Scale for Kinesiophobia (TSK) - Time necessary for completion: 10 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire is used to evaluate fear of movement and fear of (re)injury on a 4-point Likert scale ranging from "strongly disagree" to "strongly agree". Items 4, 8, 12 and 16 are inversely phrased. A higher score indicates higher levels of kinesiophobia.
Tampa Scale for Kinesiophobia (TSK) - Time necessary for completion: 10 min | T2: POST (After completing the 12-week protocol at home)
  This questionnaire is used to evaluate fear of movement and fear of (re)injury on a 4-point Likert scale ranging from "strongly disagree" to "strongly agree". Items 4, 8, 12 and 16 are inversely phrased. A higher score indicates higher levels of kinesiophobia.
Tampa Scale for Kinesiophobia (TSK) - Time necessary for completion: 10 min | T3: POST (6 months follow-up)
  This questionnaire is used to evaluate fear of movement and fear of (re)injury on a 4-point Likert scale ranging from "strongly disagree" to "strongly agree". Items 4, 8, 12 and 16 are inversely phrased. A higher score indicates higher levels of kinesiophobia.
Tampa Scale for Kinesiophobia (TSK) - Time necessary for completion: 10 min | T4: POST (18 months follow-up)
  This questionnaire is used to evaluate fear of movement and fear of (re)injury on a 4-point Likert scale ranging from "strongly disagree" to "strongly agree". Items 4, 8, 12 and 16 are inversely phrased. A higher score indicates higher levels of kinesiophobia.
Fear-Avoidance Components Scale (FACS) - Time necessary for completion: 10 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  This questionnaire is used to evaluate fear avoidance in patients with painful medical conditions. Each item is scored on a 6-point Likert scale, resulting in scores ranging from zero ("completely disagree") to five ("completely agree"). There is a maximum total score of 100, with higher scores indicating more fear-avoidance. Five severity levels have been proposed: subclinical (0-20), mild (21-40), moderate (41- 60), severe (61-80), and extreme (81-100). The FACS-D has good reliability and validity in persons with chronic musculoskeletal pain
Fear-Avoidance Components Scale (FACS) - Time necessary for completion: 10 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire is used to evaluate fear avoidance in patients with painful medical conditions. Each item is scored on a 6-point Likert scale, resulting in scores ranging from zero ("completely disagree") to five ("completely agree"). There is a maximum total score of 100, with higher scores indicating more fear-avoidance. Five severity levels have been proposed: subclinical (0-20), mild (21-40), moderate (41- 60), severe (61-80), and extreme (81-100). The FACS-D has good reliability and validity in persons with chronic musculoskeletal pain
Fear-Avoidance Components Scale (FACS) - Time necessary for completion: 10 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire is used to evaluate fear avoidance in patients with painful medical conditions. Each item is scored on a 6-point Likert scale, resulting in scores ranging from zero ("completely disagree") to five ("completely agree"). There is a maximum total score of 100, with higher scores indicating more fear-avoidance. Five severity levels have been proposed: subclinical (0-20), mild (21-40), moderate (41- 60), severe (61-80), and extreme (81-100). The FACS-D has good reliability and validity in persons with chronic musculoskeletal pain
Fear-Avoidance Components Scale (FACS) - Time necessary for completion: 10 min | T2: POST (After completing the 12-week protocol at home)
  This questionnaire is used to evaluate fear avoidance in patients with painful medical conditions. Each item is scored on a 6-point Likert scale, resulting in scores ranging from zero ("completely disagree") to five ("completely agree"). There is a maximum total score of 100, with higher scores indicating more fear-avoidance. Five severity levels have been proposed: subclinical (0-20), mild (21-40), moderate (41- 60), severe (61-80), and extreme (81-100). The FACS-D has good reliability and validity in persons with chronic musculoskeletal pain
Fear-Avoidance Components Scale (FACS) - Time necessary for completion: 10 min | T3: POST (6 months follow-up)
  This questionnaire is used to evaluate fear avoidance in patients with painful medical conditions. Each item is scored on a 6-point Likert scale, resulting in scores ranging from zero ("completely disagree") to five ("completely agree"). There is a maximum total score of 100, with higher scores indicating more fear-avoidance. Five severity levels have been proposed: subclinical (0-20), mild (21-40), moderate (41- 60), severe (61-80), and extreme (81-100). The FACS-D has good reliability and validity in persons with chronic musculoskeletal pain
Fear-Avoidance Components Scale (FACS) - Time necessary for completion: 10 min | T4: POST (18 months follow-up)
  This questionnaire is used to evaluate fear avoidance in patients with painful medical conditions. Each item is scored on a 6-point Likert scale, resulting in scores ranging from zero ("completely disagree") to five ("completely agree"). There is a maximum total score of 100, with higher scores indicating more fear-avoidance. Five severity levels have been proposed: subclinical (0-20), mild (21-40), moderate (41- 60), severe (61-80), and extreme (81-100). The FACS-D has good reliability and validity in persons with chronic musculoskeletal pain
Self-Efficacy for Exercise (SEE) - Time necessary for completion: 5 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  This questionnaire is used to evaluate self-efficacy expectations related to the ability to continue exercising in the face of barriers to exercise. A higher score indicates higher self-efficacy for exercise.
Self-Efficacy for Exercise (SEE) - Time necessary for completion: 5 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire is used to evaluate self-efficacy expectations related to the ability to continue exercising in the face of barriers to exercise. A higher score indicates higher self-efficacy for exercise.
Self-Efficacy for Exercise (SEE) - Time necessary for completion: 5 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire is used to evaluate self-efficacy expectations related to the ability to continue exercising in the face of barriers to exercise. A higher score indicates higher self-efficacy for exercise.
Self-Efficacy for Exercise (SEE) - Time necessary for completion: 5 min | T2: POST (After completing the 12-week protocol at home)
  This questionnaire is used to evaluate self-efficacy expectations related to the ability to continue exercising in the face of barriers to exercise. A higher score indicates higher self-efficacy for exercise.
Self-Efficacy for Exercise (SEE) - Time necessary for completion: 5 min | T3: POST (6 months follow-up)
  This questionnaire is used to evaluate self-efficacy expectations related to the ability to continue exercising in the face of barriers to exercise. A higher score indicates higher self-efficacy for exercise.
Self-Efficacy for Exercise (SEE) - Time necessary for completion: 5 min | T4: POST (18 months follow-up)
  This questionnaire is used to evaluate self-efficacy expectations related to the ability to continue exercising in the face of barriers to exercise. A higher score indicates higher self-efficacy for exercise.
Expectation to recover (ETR) - Time necessary for completion: 1 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  This nominal scales is used to evaluate treatment expectation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no succes' and ten means 'very good recovery'.
Expectation to recover (ETR) - Time necessary for completion: 1 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This nominal scales is used to evaluate treatment expectation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no succes' and ten means 'very good recovery'.
Expectation to recover (ETR) - Time necessary for completion: 1 min | T1: MID (After completing the 12-week protocol in hospital)
  This nominal scales is used to evaluate treatment expectation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no succes' and ten means 'very good recovery'.
Expectation to recover (ETR) - Time necessary for completion: 1 min | T2: POST (After completing the 12-week protocol at home)
  This nominal scales is used to evaluate treatment expectation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no succes' and ten means 'very good recovery'.
Expectation to recover (ETR) - Time necessary for completion: 1 min | T3: POST (6 months follow-up)
  This nominal scales is used to evaluate treatment expectation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no succes' and ten means 'very good recovery'.
Expectation to recover (ETR) - Time necessary for completion: 1 min | T4: POST (18 months follow-up)
  This nominal scales is used to evaluate treatment expectation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no succes' and ten means 'very good recovery'.
Brief Illness Perception Questionnaire (b-IPQ) - Time necessary for completion: 5 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  This questionnaire is used to evaluate cognitive and emotional representations of illness. The Brief IPQ uses a single-item scale approach to assess perception on a 0-10 response scale. . A higher score indicates more negative perceptions.
Brief Illness Perception Questionnaire (b-IPQ) - Time necessary for completion: 5 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire is used to evaluate cognitive and emotional representations of illness. The Brief IPQ uses a single-item scale approach to assess perception on a 0-10 response scale. . A higher score indicates more negative perceptions.
Brief Illness Perception Questionnaire (b-IPQ) - Time necessary for completion: 5 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire is used to evaluate cognitive and emotional representations of illness. The Brief IPQ uses a single-item scale approach to assess perception on a 0-10 response scale. . A higher score indicates more negative perceptions.
Brief Illness Perception Questionnaire (b-IPQ) - Time necessary for completion: 5 min | T2: POST (After completing the 12-week protocol at home)
  This questionnaire is used to evaluate cognitive and emotional representations of illness. The Brief IPQ uses a single-item scale approach to assess perception on a 0-10 response scale. . A higher score indicates more negative perceptions.
Brief Illness Perception Questionnaire (b-IPQ) - Time necessary for completion: 5 min | T3: POST (6 months follow-up)
  This questionnaire is used to evaluate cognitive and emotional representations of illness. The Brief IPQ uses a single-item scale approach to assess perception on a 0-10 response scale. . A higher score indicates more negative perceptions.
Brief Illness Perception Questionnaire (b-IPQ) - Time necessary for completion: 5 min | T4: POST (18 months follow-up)
  This questionnaire is used to evaluate cognitive and emotional representations of illness. The Brief IPQ uses a single-item scale approach to assess perception on a 0-10 response scale. . A higher score indicates more negative perceptions.
Injustice Experience Questionnaire (IEQ) - Time necessary for completion: 5 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  This questionnaire is used to evaluate perceived injustice and consists of of 12 items, scored on a range from zero "not at all" to four "all the time". Higher total scores reflect higher levels of perceived injustice. Cut-off scores of 19 and 30 are reported for medium and high levels of perceived injustice, respectively.
Injustice Experience Questionnaire (IEQ) - Time necessary for completion: 5 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire is used to evaluate perceived injustice and consists of of 12 items, scored on a range from zero "not at all" to four "all the time". Higher total scores reflect higher levels of perceived injustice. Cut-off scores of 19 and 30 are reported for medium and high levels of perceived injustice, respectively.
Injustice Experience Questionnaire (IEQ) - Time necessary for completion: 5 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire is used to evaluate perceived injustice and consists of of 12 items, scored on a range from zero "not at all" to four "all the time". Higher total scores reflect higher levels of perceived injustice. Cut-off scores of 19 and 30 are reported for medium and high levels of perceived injustice, respectively.
Injustice Experience Questionnaire (IEQ) - Time necessary for completion: 5 min | T2: POST (After completing the 12-week protocol at home)
  This questionnaire is used to evaluate perceived injustice and consists of of 12 items, scored on a range from zero "not at all" to four "all the time". Higher total scores reflect higher levels of perceived injustice. Cut-off scores of 19 and 30 are reported for medium and high levels of perceived injustice, respectively.
Injustice Experience Questionnaire (IEQ) - Time necessary for completion: 5 min | T3: POST (6 months follow-up)
  This questionnaire is used to evaluate perceived injustice and consists of of 12 items, scored on a range from zero "not at all" to four "all the time". Higher total scores reflect higher levels of perceived injustice. Cut-off scores of 19 and 30 are reported for medium and high levels of perceived injustice, respectively.
Injustice Experience Questionnaire (IEQ) - Time necessary for completion: 5 min | T4: POST (18 months follow-up)
  This questionnaire is used to evaluate perceived injustice and consists of of 12 items, scored on a range from zero "not at all" to four "all the time". Higher total scores reflect higher levels of perceived injustice. Cut-off scores of 19 and 30 are reported for medium and high levels of perceived injustice, respectively.
A maximal cardiopulmonary exercise test - Time necessary for completion: 30 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  A bicycle ergometer (eBike Basic, General Electric GmbH, Bitz, Germany) with pulmonary gas exchange analysis (MetaMax 3B, Cortex Biophysik GmbH, Leipzig, Germany) will be used. Herein, a low workload gradually increases each minute (30W+15W/min). Maximal oxygen uptake (VO2max) and maximal workload through cycling time (min.) are evaluated through breath-by-breath gas exchange analysis and heartrate monitoring (H10, Polar Electro). A minimum respiratory exchange ratio (RER) threshold of 1.10 is used to evaluate proper validity of the maximum effort.
A maximal cardiopulmonary exercise test - Time necessary for completion: 30 min | T1: MID (After completing the 12-week protocol in hospital)
  A bicycle ergometer (eBike Basic, General Electric GmbH, Bitz, Germany) with pulmonary gas exchange analysis (MetaMax 3B, Cortex Biophysik GmbH, Leipzig, Germany) will be used. Herein, a low workload gradually increases each minute (30W+15W/min). Maximal oxygen uptake (VO2max) and maximal workload through cycling time (min.) are evaluated through breath-by-breath gas exchange analysis and heartrate monitoring (H10, Polar Electro). A minimum respiratory exchange ratio (RER) threshold of 1.10 is used to evaluate proper validity of the maximum effort.
A maximal cardiopulmonary exercise test - Time necessary for completion: 30 min | T2: POST (After completing the 12-week protocol at home)
  A bicycle ergometer (eBike Basic, General Electric GmbH, Bitz, Germany) with pulmonary gas exchange analysis (MetaMax 3B, Cortex Biophysik GmbH, Leipzig, Germany) will be used. Herein, a low workload gradually increases each minute (30W+15W/min). Maximal oxygen uptake (VO2max) and maximal workload through cycling time (min.) are evaluated through breath-by-breath gas exchange analysis and heartrate monitoring (H10, Polar Electro). A minimum respiratory exchange ratio (RER) threshold of 1.10 is used to evaluate proper validity of the maximum effort.
A maximal cardiopulmonary exercise test - Time necessary for completion: 30 min | T3: POST (6 months follow-up)
  A bicycle ergometer (eBike Basic, General Electric GmbH, Bitz, Germany) with pulmonary gas exchange analysis (MetaMax 3B, Cortex Biophysik GmbH, Leipzig, Germany) will be used. Herein, a low workload gradually increases each minute (30W+15W/min). Maximal oxygen uptake (VO2max) and maximal workload through cycling time (min.) are evaluated through breath-by-breath gas exchange analysis and heartrate monitoring (H10, Polar Electro). A minimum respiratory exchange ratio (RER) threshold of 1.10 is used to evaluate proper validity of the maximum effort.
A maximal cardiopulmonary exercise test - Time necessary for completion: 30 min | T4: POST (18 months follow-up)
  A bicycle ergometer (eBike Basic, General Electric GmbH, Bitz, Germany) with pulmonary gas exchange analysis (MetaMax 3B, Cortex Biophysik GmbH, Leipzig, Germany) will be used. Herein, a low workload gradually increases each minute (30W+15W/min). Maximal oxygen uptake (VO2max) and maximal workload through cycling time (min.) are evaluated through breath-by-breath gas exchange analysis and heartrate monitoring (H10, Polar Electro). A minimum respiratory exchange ratio (RER) threshold of 1.10 is used to evaluate proper validity of the maximum effort.
International Physical Activity Questionnaire short form (IPAQ-sf) - Time necessary for completion: 5 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire is used to estimate physical activity level. The questionnaire consists of 7 questions. A higher score corresponds to a more physically demanding activity level. This questionnaire is reliable and valid for use in persons with chronic low back pain.
International Physical Activity Questionnaire short form (IPAQ-sf) - Time necessary for completion: 5 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire is used to estimate physical activity level. The questionnaire consists of 7 questions. A higher score corresponds to a more physically demanding activity level. This questionnaire is reliable and valid for use in persons with chronic low back pain.
International Physical Activity Questionnaire short form (IPAQ-sf) - Time necessary for completion: 5 min | T2: POST (6 months follow-up)
  This questionnaire is used to estimate physical activity level. The questionnaire consists of 7 questions. A higher score corresponds to a more physically demanding activity level. This questionnaire is reliable and valid for use in persons with chronic low back pain.
International Physical Activity Questionnaire short form (IPAQ-sf) - Time necessary for completion: 5 min | T3: POST (18 months follow-up)
  This questionnaire is used to estimate physical activity level. The questionnaire consists of 7 questions. A higher score corresponds to a more physically demanding activity level. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Pittsburg Sleep Quality Index (PSQI) - Time necessary for completion: 10 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire (19 items, three-point scale) evaluates last month's sleep quality in seven domains: sleep latency time, sleep duration, sleep medication, daytime functioning, sleep-related problems
Pittsburg Sleep Quality Index (PSQI) - Time necessary for completion: 10 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire (19 items, three-point scale) evaluates last month's sleep quality in seven domains: sleep latency time, sleep duration, sleep medication, daytime functioning, sleep-related problems
Pittsburg Sleep Quality Index (PSQI) - Time necessary for completion: 10 min | T2: POST (After completing the 12-week protocol at home)
  This questionnaire (19 items, three-point scale) evaluates last month's sleep quality in seven domains: sleep latency time, sleep duration, sleep medication, daytime functioning, sleep-related problems
Pittsburg Sleep Quality Index (PSQI) - Time necessary for completion: 10 min | T3: POST (6 months follow-up)
  This questionnaire (19 items, three-point scale) evaluates last month's sleep quality in seven domains: sleep latency time, sleep duration, sleep medication, daytime functioning, sleep-related problems
Pittsburg Sleep Quality Index (PSQI) - Time necessary for completion: 10 min | T4: POST (18 months follow-up)
  This questionnaire (19 items, three-point scale) evaluates last month's sleep quality in seven domains: sleep latency time, sleep duration, sleep medication, daytime functioning, sleep-related problems
Heart rate variability (HRV) - Time necessary for completion: 20 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  To evaluate cardiac autonomic function, HRV will be measured. Patients are guided to a quiet low stimulus room and instructed to remain in a supine position for 7 min before beat-to-beat intervals (R-R) are registered using a validated heart rate band (H10, Polar Electro) synchronized with a heart rate monitor (Ignite, Polar Electro). RR data will be extracted using Polar Flow software. The first two minutes are not included to guarantee a steady heart rate. Artefact correction is set at very low. Raw RR data will be analysed with HRV software (Kubios HRV, Kubios Oy) and includes time domain analysis, frequency domain analysis, nonlinear analysis, and time- frequency analysis.
Heart rate variability (HRV) - Time necessary for completion: 20 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  To evaluate cardiac autonomic function, HRV will be measured. Patients are guided to a quiet low stimulus room and instructed to remain in a supine position for 7 min before beat-to-beat intervals (R-R) are registered using a validated heart rate band (H10, Polar Electro) synchronized with a heart rate monitor (Ignite, Polar Electro). RR data will be extracted using Polar Flow software. The first two minutes are not included to guarantee a steady heart rate. Artefact correction is set at very low. Raw RR data will be analysed with HRV software (Kubios HRV, Kubios Oy) and includes time domain analysis, frequency domain analysis, nonlinear analysis, and time- frequency analysis.
Heart rate variability (HRV) - Time necessary for completion: 20 min | T1: MID (After completing the 12-week protocol in hospital)
  To evaluate cardiac autonomic function, HRV will be measured. Patients are guided to a quiet low stimulus room and instructed to remain in a supine position for 7 min before beat-to-beat intervals (R-R) are registered using a validated heart rate band (H10, Polar Electro) synchronized with a heart rate monitor (Ignite, Polar Electro). RR data will be extracted using Polar Flow software. The first two minutes are not included to guarantee a steady heart rate. Artefact correction is set at very low. Raw RR data will be analysed with HRV software (Kubios HRV, Kubios Oy) and includes time domain analysis, frequency domain analysis, nonlinear analysis, and time- frequency analysis.
Heart rate variability (HRV) - Time necessary for completion: 20 min | T2: POST (After completing the 12-week protocol at home)
  To evaluate cardiac autonomic function, HRV will be measured. Patients are guided to a quiet low stimulus room and instructed to remain in a supine position for 7 min before beat-to-beat intervals (R-R) are registered using a validated heart rate band (H10, Polar Electro) synchronized with a heart rate monitor (Ignite, Polar Electro). RR data will be extracted using Polar Flow software. The first two minutes are not included to guarantee a steady heart rate. Artefact correction is set at very low. Raw RR data will be analysed with HRV software (Kubios HRV, Kubios Oy) and includes time domain analysis, frequency domain analysis, nonlinear analysis, and time- frequency analysis.
Heart rate variability (HRV) - Time necessary for completion: 20 min | T3: POST (6 months follow-up)
  To evaluate cardiac autonomic function, HRV will be measured. Patients are guided to a quiet low stimulus room and instructed to remain in a supine position for 7 min before beat-to-beat intervals (R-R) are registered using a validated heart rate band (H10, Polar Electro) synchronized with a heart rate monitor (Ignite, Polar Electro). RR data will be extracted using Polar Flow software. The first two minutes are not included to guarantee a steady heart rate. Artefact correction is set at very low. Raw RR data will be analysed with HRV software (Kubios HRV, Kubios Oy) and includes time domain analysis, frequency domain analysis, nonlinear analysis, and time- frequency analysis.
Heart rate variability (HRV) - Time necessary for completion: 20 min | T4: POST (18 months follow-up)
  To evaluate cardiac autonomic function, HRV will be measured. Patients are guided to a quiet low stimulus room and instructed to remain in a supine position for 7 min before beat-to-beat intervals (R-R) are registered using a validated heart rate band (H10, Polar Electro) synchronized with a heart rate monitor (Ignite, Polar Electro). RR data will be extracted using Polar Flow software. The first two minutes are not included to guarantee a steady heart rate. Artefact correction is set at very low. Raw RR data will be analysed with HRV software (Kubios HRV, Kubios Oy) and includes time domain analysis, frequency domain analysis, nonlinear analysis, and time- frequency analysis.
The EuroQoL EQ-5D - Time necessary for completion: 10 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire is used to evaluate to collect health-related Quality of Life (QoL). This validated Dutch questionnaire measures QoL using five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A high score corresponds to a better QOL.
The EuroQoL EQ-5D - Time necessary for completion: 10 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire is used to evaluate to collect health-related Quality of Life (QoL). This validated Dutch questionnaire measures QoL using five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A high score corresponds to a better QOL.
The EuroQoL EQ-5D - Time necessary for completion: 10 min | T2: POST (After completing the 12-week protocol at home)
  This questionnaire is used to evaluate to collect health-related Quality of Life (QoL). This validated Dutch questionnaire measures QoL using five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A high score corresponds to a better QOL.
The EuroQoL EQ-5D - Time necessary for completion: 10 min | T3: POST (6 months follow-up)
  This questionnaire is used to evaluate to collect health-related Quality of Life (QoL). This validated Dutch questionnaire measures QoL using five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A high score corresponds to a better QOL.
The EuroQoL EQ-5D - Time necessary for completion: 10 min | T4: POST (18 months follow-up)
  This questionnaire is used to evaluate to collect health-related Quality of Life (QoL). This validated Dutch questionnaire measures QoL using five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A high score corresponds to a better QOL.
The number of completed therapy sessions - Time necessary for completion: 1 min | T1: MID (After completing the 12-week protocol in hospital)
  The number of completed therapy sessions within the protocol will be registered during the execution of the intervention (at the hospital and at home). Reasons for non-adherence will be inventoried.
The number of completed therapy sessions - Time necessary for completion: 1 min | T2: POST (After completing the 12-week protocol at home)
  The number of completed therapy sessions within the protocol will be registered during the execution of the intervention (at the hospital and at home). Reasons for non-adherence will be inventoried.
The number of completed therapy sessions - Time necessary for completion: 1 min | T3: POST (6 months follow-up)
  The number of completed therapy sessions within the protocol will be registered during the execution of the intervention (at the hospital and at home). Reasons for non-adherence will be inventoried.
The number of completed therapy sessions - Time necessary for completion: 1 min | T4: POST (18 months follow-up)
  The number of completed therapy sessions within the protocol will be registered during the execution of the intervention (at the hospital and at home). Reasons for non-adherence will be inventoried.
Exercise adherence rating Scale (EARS) - Time necessary for completion: 10 min | T1: MID (After completing the 12-week protocol in hospital)
  The adherence to prescribed home exercises will be assessed using EARS, a 16-item questionnaire. A higher score indicates higher adherence.
Exercise adherence rating Scale (EARS) - Time necessary for completion: 10 min | T2: POST (After completing the 12-week protocol at home)
  The adherence to prescribed home exercises will be assessed using EARS, a 16-item questionnaire. A higher score indicates higher adherence.
Exercise adherence rating Scale (EARS) - Time necessary for completion: 10 min | T3: POST (6 months follow-up)
  The adherence to prescribed home exercises will be assessed using EARS, a 16-item questionnaire. A higher score indicates higher adherence.
Exercise adherence rating Scale (EARS) - Time necessary for completion: 10 min | T4: POST (18 months follow-up)
  The adherence to prescribed home exercises will be assessed using EARS, a 16-item questionnaire. A higher score indicates higher adherence.
System Usability Scale (SUS) - Time necessary for completion: 5 min | T2: POST (After completing the 12-week protocol at home)
  Participants will complete this questionnaire to assess perceived usability of the smartphone application. SUS is a standard 10-item questionnaire in which responses are measured on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Questions 1, 3, 5, 7, and 9 are positive and questions 2, 4, 6, 8, and 10 are negative. A total SUS score is derived by summing the individual scores and multiplying by 2.5, which yields a score ranging between 0 (worst) and 100 (absolute best). A score >68 is considered above average usability and >80 considered high usability and a level at which participants are likely to recommend the product to peers.
System Usability Scale (SUS) - Time necessary for completion: 5 min | T3: POST (6 months follow-up)
  Participants will complete this questionnaire to assess perceived usability of the smartphone application. SUS is a standard 10-item questionnaire in which responses are measured on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Questions 1, 3, 5, 7, and 9 are positive and questions 2, 4, 6, 8, and 10 are negative. A total SUS score is derived by summing the individual scores and multiplying by 2.5, which yields a score ranging between 0 (worst) and 100 (absolute best). A score >68 is considered above average usability and >80 considered high usability and a level at which participants are likely to recommend the product to peers.
System Usability Scale (SUS) - Time necessary for completion: 5 min | T4: POST (18 months follow-up)
  Participants will complete this questionnaire to assess perceived usability of the smartphone application. SUS is a standard 10-item questionnaire in which responses are measured on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Questions 1, 3, 5, 7, and 9 are positive and questions 2, 4, 6, 8, and 10 are negative. A total SUS score is derived by summing the individual scores and multiplying by 2.5, which yields a score ranging between 0 (worst) and 100 (absolute best). A score >68 is considered above average usability and >80 considered high usability and a level at which participants are likely to recommend the product to peers.
User Version of the Mobile Application Rating Scale (uMARS)- Time necessary for completion: 5 min | T2: POST (After completing the 12-week protocol at home)
  The uMARS is a a 20-item questionnaire that includes 4 objective quality subscales: engagement, functionality, aesthetics, and information quality, and 1 subjective quality subscale. Each item is scored on a 5-point Likert scale. Both individual items aswell as a mean overall score can be used for evaluation.
User Version of the Mobile Application Rating Scale (uMARS)- Time necessary for completion: 5 min | T3: POST (6 months follow-up)
  The uMARS is a a 20-item questionnaire that includes 4 objective quality subscales: engagement, functionality, aesthetics, and information quality, and 1 subjective quality subscale. Each item is scored on a 5-point Likert scale. Both individual items aswell as a mean overall score can be used for evaluation.
User Version of the Mobile Application Rating Scale (uMARS)- Time necessary for completion: 5 min | T4: POST (18 months follow-up)
  The uMARS is a a 20-item questionnaire that includes 4 objective quality subscales: engagement, functionality, aesthetics, and information quality, and 1 subjective quality subscale. Each item is scored on a 5-point Likert scale. Both individual items aswell as a mean overall score can be used for evaluation.
Intrinsic Motivation Inventory (IMI) - Time necessary for completion: 10 min | T2: POST (After completing the 12-week protocol at home)
  This is a nominal 35 item questionnaire that assesses the multidimensional subjective experience while performing a certain activity yielding six subscales (interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, and perceived choice), with the possibility of independent scoring for each scale and a general scoring. A higher score correlates to higher intrinsic motivation (total range 35-245).
Intrinsic Motivation Inventory (IMI) - Time necessary for completion: 10 min | T3: POST (6 months follow-up)
  This is a nominal 35 item questionnaire that assesses the multidimensional subjective experience while performing a certain activity yielding six subscales (interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, and perceived choice), with the possibility of independent scoring for each scale and a general scoring. A higher score correlates to higher intrinsic motivation (total range 35-245).
Intrinsic Motivation Inventory (IMI) - Time necessary for completion: 10 min | T4: POST (18 months follow-up)
  This is a nominal 35 item questionnaire that assesses the multidimensional subjective experience while performing a certain activity yielding six subscales (interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, and perceived choice), with the possibility of independent scoring for each scale and a general scoring. A higher score correlates to higher intrinsic motivation (total range 35-245).
iMTA Productivity Cost Questionnaire (iPCQ) - Time necessary for completion: 15 min | T1: MID (After completing the 12-week protocol in hospital)
  absenteeism at work/loss of productivity will be evaluated using the IPCQ. iPCQ includes three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presentism, and 3) productivity losses due to unpaid work. iPCQ delivers necessary input to calculate costs associated to productivity loss using the Human Capital Approach for short-term absence and Friction Cost Method for long-term absence. The HCA values the time during the whole period of work inability due to sick leave by multiplying total number of days of work absenteeism by national average labor costs per day. FCM calculates the value of productivity loss by multiplying national labor costs per day by the friction period (i.e. time span to restore initial production level after an employee becomes absent from work). In accordance with KCE guidelines, informal home care (i.e. care by relatives and family) and unpaid work will be measured, but not valued.
iMTA Productivity Cost Questionnaire (iPCQ) - Time necessary for completion: 15 min | T2: POST (After completing the 12-week protocol at home)
  absenteeism at work/loss of productivity will be evaluated using the IPCQ. iPCQ includes three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presentism, and 3) productivity losses due to unpaid work. iPCQ delivers necessary input to calculate costs associated to productivity loss using the Human Capital Approach for short-term absence and Friction Cost Method for long-term absence. The HCA values the time during the whole period of work inability due to sick leave by multiplying total number of days of work absenteeism by national average labor costs per day. FCM calculates the value of productivity loss by multiplying national labor costs per day by the friction period (i.e. time span to restore initial production level after an employee becomes absent from work). In accordance with KCE guidelines, informal home care (i.e. care by relatives and family) and unpaid work will be measured, but not valued.
iMTA Productivity Cost Questionnaire (iPCQ) - Time necessary for completion: 15 min | T3: POST (6 months follow-up)
  absenteeism at work/loss of productivity will be evaluated using the IPCQ. iPCQ includes three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presentism, and 3) productivity losses due to unpaid work. iPCQ delivers necessary input to calculate costs associated to productivity loss using the Human Capital Approach for short-term absence and Friction Cost Method for long-term absence. The HCA values the time during the whole period of work inability due to sick leave by multiplying total number of days of work absenteeism by national average labor costs per day. FCM calculates the value of productivity loss by multiplying national labor costs per day by the friction period (i.e. time span to restore initial production level after an employee becomes absent from work). In accordance with KCE guidelines, informal home care (i.e. care by relatives and family) and unpaid work will be measured, but not valued.
iMTA Productivity Cost Questionnaire (iPCQ) - Time necessary for completion: 15 min | T4: POST (18 months follow-up)
  absenteeism at work/loss of productivity will be evaluated using the IPCQ. iPCQ includes three modules measuring productivity losses of paid work due to 1) absenteeism and 2) presentism, and 3) productivity losses due to unpaid work. iPCQ delivers necessary input to calculate costs associated to productivity loss using the Human Capital Approach for short-term absence and Friction Cost Method for long-term absence. The HCA values the time during the whole period of work inability due to sick leave by multiplying total number of days of work absenteeism by national average labor costs per day. FCM calculates the value of productivity loss by multiplying national labor costs per day by the friction period (i.e. time span to restore initial production level after an employee becomes absent from work). In accordance with KCE guidelines, informal home care (i.e. care by relatives and family) and unpaid work will be measured, but not valued.
In-hospital costs - Time necessary for completion: 5 min | T1: MID (After completing the 12-week protocol in hospital)
  The in-hospital costs of participants will be calculated using accounting records of the participating hospitals, which are highly comparable since both use a standardized program in each of the three groups. Most important in-hospital cost categories are: rehabilitation, medication and devices, consultation fees, staff fees, surgeries. This list is however not exhaustive. The hospitals' accounting information will give more insight in the interventions and medication given to participants.
In-hospital costs - Time necessary for completion: 5 min | T2: POST (After completing the 12-week protocol at home)
  The in-hospital costs of participants will be calculated using accounting records of the participating hospitals, which are highly comparable since both use a standardized program in each of the three groups. Most important in-hospital cost categories are: rehabilitation, medication and devices, consultation fees, staff fees, surgeries. This list is however not exhaustive. The hospitals' accounting information will give more insight in the interventions and medication given to participants.
In-hospital costs - Time necessary for completion: 5 min | T3: POST (6 months follow-up)
  The in-hospital costs of participants will be calculated using accounting records of the participating hospitals, which are highly comparable since both use a standardized program in each of the three groups. Most important in-hospital cost categories are: rehabilitation, medication and devices, consultation fees, staff fees, surgeries. This list is however not exhaustive. The hospitals' accounting information will give more insight in the interventions and medication given to participants.
In-hospital costs - Time necessary for completion: 5 min | T4: POST (18 months follow-up)
  The in-hospital costs of participants will be calculated using accounting records of the participating hospitals, which are highly comparable since both use a standardized program in each of the three groups. Most important in-hospital cost categories are: rehabilitation, medication and devices, consultation fees, staff fees, surgeries. This list is however not exhaustive. The hospitals' accounting information will give more insight in the interventions and medication given to participants.
Healthcare utilization costs - Time necessary for completion: 5 min | T3: POST (6 months follow-up)
  a self-reported healthcare utilization questionnaire will be used by PEC-UH to measure the out-of-hospital healthcare utilization and costs (additional, extramural medical interventions and medication related to CLBP).
Healthcare utilization costs - Time necessary for completion: 5 min | T4: POST (18 months follow-up)
  a self-reported healthcare utilization questionnaire will be used by PEC-UH to measure the out-of-hospital healthcare utilization and costs (additional, extramural medical interventions and medication related to CLBP).
C-reactive protein (CRP) testing - Time necessary for completion: 2 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  A non-invasive finger-prick blood sampling technique will quantify CRP levels using the QuickRead Go by Aidian, Finland.
C-reactive protein (CRP) testing - Time necessary for completion: 2 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  A non-invasive finger-prick blood sampling technique will quantify CRP levels using the QuickRead Go by Aidian, Finland.
C-reactive protein (CRP) testing - Time necessary for completion: 2 min | T1: MID (After completing the 12-week protocol in hospital)
  A non-invasive finger-prick blood sampling technique will quantify CRP levels using the QuickRead Go by Aidian, Finland.
C-reactive protein (CRP) testing - Time necessary for completion: 2 min | T2: POST (After completing the 12-week protocol at home)
  A non-invasive finger-prick blood sampling technique will quantify CRP levels using the QuickRead Go by Aidian, Finland.
C-reactive protein (CRP) testing - Time necessary for completion: 2 min | T3: POST (6 months follow-up)
  A non-invasive finger-prick blood sampling technique will quantify CRP levels using the QuickRead Go by Aidian, Finland.
C-reactive protein (CRP) testing - Time necessary for completion: 2 min | T4: POST (18 months follow-up)
  A non-invasive finger-prick blood sampling technique will quantify CRP levels using the QuickRead Go by Aidian, Finland.
Hemoglobin A1c (HbA1c) testing - Time necessary for completion: 2 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  A non-invasive finger-prick blood sampling technique will quantify glucose concentration in the bloodstream using the QuickRead Go by Aidian, Finland.
Hemoglobin A1c (HbA1c) testing - Time necessary for completion: 2 min | T1: MID (After completing the 12-week protocol in hospital)
  A non-invasive finger-prick blood sampling technique will quantify glucose concentration in the bloodstream using the QuickRead Go by Aidian, Finland.
Hemoglobin A1c (HbA1c) testing - Time necessary for completion: 2 min | T2: POST (After completing the 12-week protocol at home)
  A non-invasive finger-prick blood sampling technique will quantify glucose concentration in the bloodstream using the QuickRead Go by Aidian, Finland.
Hemoglobin A1c (HbA1c) testing - Time necessary for completion: 2 min | T3: POST (6 months follow-up)
  A non-invasive finger-prick blood sampling technique will quantify glucose concentration in the bloodstream using the QuickRead Go by Aidian, Finland.
Hemoglobin A1c (HbA1c) testing - Time necessary for completion: 2 min | T4: POST (18 months follow-up)
  A non-invasive finger-prick blood sampling technique will quantify glucose concentration in the bloodstream using the QuickRead Go by Aidian, Finland.
Positive and Negative Affect Schedule (PANAS) - Time necessary for completion: 5 min | T-1: PRE (pre biopsychosocial education program, 2 weeks before the start of intervention)
  This questionnaire is used to evaluate participants' emotional states and fluctuations on a 5-point Likert scale and consists of 10 items representing positive affect dimensions and 10 items representing negative affect dimensions.
Positive and Negative Affect Schedule (PANAS) - Time necessary for completion: 5 min | T0: PRE (post biopsychosocial education program, at the start of intervention)
  This questionnaire is used to evaluate participants' emotional states and fluctuations on a 5-point Likert scale and consists of 10 items representing positive affect dimensions and 10 items representing negative affect dimensions.
Positive and Negative Affect Schedule (PANAS) - Time necessary for completion: 5 min | T1: MID (After completing the 12-week protocol in hospital)
  This questionnaire is used to evaluate participants' emotional states and fluctuations on a 5-point Likert scale and consists of 10 items representing positive affect dimensions and 10 items representing negative affect dimensions.
Positive and Negative Affect Schedule (PANAS) - Time necessary for completion: 5 min | T2: POST (After completing the 12-week protocol at home)
  This questionnaire is used to evaluate participants' emotional states and fluctuations on a 5-point Likert scale and consists of 10 items representing positive affect dimensions and 10 items representing negative affect dimensions.
Positive and Negative Affect Schedule (PANAS) - Time necessary for completion: 5 min | T3: POST (6 months follow-up)
  This questionnaire is used to evaluate participants' emotional states and fluctuations on a 5-point Likert scale and consists of 10 items representing positive affect dimensions and 10 items representing negative affect dimensions.
Positive and Negative Affect Schedule (PANAS) - Time necessary for completion: 5 min | T4: POST (18 months follow-up)
  This questionnaire is used to evaluate participants' emotional states and fluctuations on a 5-point Likert scale and consists of 10 items representing positive affect dimensions and 10 items representing negative affect dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Annick Timmermans, Principal Investigator — Hasselt University
Locations (4):
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen (UZA), Wilrijk, Antwerpen
  - University of Antwerp, Wilrijk, Antwerpen
  - Hasselt University, Diepenbeek, Limburg
  - Jessa Ziekenhuis, Hasselt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Eetvelde JS, Timmermans AAA, Coninx K, Kempeneers K, Meeus M, Marneffe W, Meus T, Meuwissen I, Roussel NA, Stassijns G, Verbrugghe J. Technology supported High Intensity Training in chronic non-specific low back pain (the Techno-HIT trial): study protocol of a randomised controlled trial. BMJ Open Sport Exerc Med. 2024 Oct 7;10(4):e002180. doi: 10.1136/bmjsem-2024-002180. eCollection 2024. PMID 39381416